CLINICAL TRIAL: NCT04897243
Title: A Prospective Cohort Study Examining Two Models of Care for B/F/TAF Initiation in HIV-infected, ART-naïve Newly Referred Patients
Brief Title: Antiretroviral Speed Access Program
Acronym: ASAP
Status: Recruiting | Type: Observational
Sponsor: Dr. Bertrand Lebouche (Other)
Responsible Party: Sponsor-Investigator, Dr. Bertrand Lebouche, Clinical Scientist and Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: IN-US-380-4670
Record Dates: First submitted 2021-04-13; First posted 2021-05-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: HIV Infection
Keywords: HIV; multidisciplinary model of care; patient-reported experience; ART initiation; patient engagement
MeSH Terms: conditions — HIV Infections; Patient Participation | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Multidisciplinary model of care: The Chronic Viral Illness Service at the Glen hospital of the MUHC will provide care with a multidisciplinary assessment, according to local current standard practice. Each newly-referred patient at the CVIS will be first received by a dedicated nurse, who then orients referral to a physician and/or a social worker and/or a pharmacist.
  Interventions: Drug: Biktarvy; Behavioral: Patient Experience
- Physician-only model of care: The Jewish General Hospital will provide care as per current local standard practice. Each newly-referred patient will be assessed by a clinician. Blood tests will be performed by central laboratory nurses who are not part of the HIV clinic.
  Interventions: Drug: Biktarvy; Behavioral: Patient Experience

INTERVENTIONS:
Drug: Biktarvy — B/F/TAF (Biktarvy®) is a fixed-dose combination of bictegravir (50 mg), emtricitabine (200 mg), and tenofovir alafenamide (25 mg), administered orally, once daily, without food requirements. Participating patients will receive the medication free of charge.
  Other Names: B/F/TAF
Behavioral: Patient Experience — To capture and integrate the patient experience, this study will collect patient-reported experience measures, conduct qualitative interviews, and engage patients as well as providers.

SUMMARY:
Migrant populations represent an increasing proportion of newly referred people living with HIV in Canada, particularly in Quebec. Timely HIV care of newly referred patients has important individual-level health benefits that can result in decreased transmission and benefit the society as a whole. Yet, the timing of events in the HIV care cascade (from linkage to care to sustained viral suppression) together with the specific experience of care of these vulnerable populations (asylum-seekers, international students, patients with no status) who often face specific psycho-social and/or financial issues, has rarely been studied. In particular, little is known about their experience of HIV care whether they are referred to a multidisciplinary clinic or a physician-only clinic.

In a context where B/F/TAF will be provided free-of-charge to all enrolled participants including migrant populations, we aim to investigate what model of care can best address current deficiencies in the standard HIV care cascade for newly-referred patients, which often involves delays in linkage to care and starting ART.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Newly referred at the study site
3. HIV-1 infected (fourth generation HIV Ag/Ab combination assay)
4. Treatment-naïve to all anti-HIV therapy, except for the use for pre-exposure prophylaxis (PrEP) or post-exposure prophylaxis (PEP), up to one month prior to screening
5. Estimated GFR >30 mL/min/1.73m2 according to the Cockcroft-Gault formula for creatinine clearance
6. Must be willing and able to understand the requirements of study participation and provide signed and dated written informed consent prior to screening
7. Female participants who are willing to use acceptable methods of birth control as defined in the protocol

Exclusion Criteria:

1. Have received anti-HIV therapy previously, except for PrEP or PEP taken up to one month prior to screening
2. Viral load <100 copies/mL, high suspicion of non-reported ART use or being a long-term nonprogressor or elite controller
3. Concomitant use of drugs with contraindication or drug-drug interactions with B/F/TAF
4. Documented historic or baseline allergy to any of the components of B/F/TAF
5. Estimated eGFR (by Cockcroft-Gault formula) < 30 mL/min
6. Pregnant, breast-feeding or planning or suspected to get pregnant
7. Involvement in any other interventional HIV studies during the study period
8. Has any reason, in the opinion of the investigator, which would make the candidate inappropriate for participation in an investigative study involving oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected patients, ART-naïve, newly referred at the study sites (CVIS or JGH). Based on experience, over 70% of these new patients would qualify as vulnerable (asylum seekers, migrants, international students with low healthcare coverage).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in perceived problem solving | Change through study completion, an average of 2 years by model of care
  Subscale of the Patient-Assessment of Chronic Illness Care (PACIC) measure. The PACIC consists of 5 scales and an overall summary score. Items 12 to 15 are about "Problem Solving/Contextual"; each can be scored from 1 to 5 (higher scores mean a better outcome and lower scores mean a worse outcome).
Change in perceived provider empathy | Change through study completion, an average of 2 years by model of care
  The Consultation and Relational Empathy (CARE) measure
Change in treatment satisfaction | Change through study completion, an average of 2 years by model of care
  HIV Treatment Satisfaction Questionnaire (HIVTSQ). The revised version of the HIVTSQ-status contains 10 items (Woodcock et al., 2006). Items are rated from 0 to 6, with response options adjusted to the item (higher scores mean a better outcome and lower scores mean a worse outcome).
Perceived unmet healthcare needs | Change through study completion, an average of 2 years by model of care
  Question taken from the Canadian Community Health Survey (CCHS 2.1)

SECONDARY OUTCOMES:
Change in self-reported adherence to ART | Change through study completion, an average of 2 years by model of care
  Self-reported ART in the past 30 days
Time to viral suppression | From weeks 1 to 96
  Time to viral suppression (i.e. less than 50 copies/ml), from treatment initiation, by model of care
Time to treatment initiation | From first clinic appointment (prior to week 1)
  Days between the first appointment at the clinic and first patient-reported dose of ART
Change in adherence to ART | Between weeks 1 and 96
  Based on pill counts each time a patient returns for refills
Change in appointment attendance | Between weeks 1 and 96
  Attendance to each scheduled study visit (+- 7 days or +- 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Lebouché, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada